CLINICAL TRIAL: NCT04159337
Title: A Prospective Study on Companion Diagnosis by NGS-based Large-panel in Targeted Drug Delivery and Immunotherapy of Lung Cancer
Brief Title: NGS-based Large-panel in Targeted Drug Delivery and Immunotherapy of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Chief physician, Shanghai Chest Hospital
Other Study IDs: ShanghaiChest0015
Record Dates: First submitted 2019-10-23; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The method of gene mutation detection — All samples were detected by large-panel, whereas some of which were also detected by WES.

SUMMARY:
Companion diagnosis by large-panel is in increasing acceptance and need during clinical cancer management. The purpose of this trial is to investigate the benefit of large-panel NGS analysis in companion diagnosis of advanced lung cancer patients and further optimize the parameters.

DETAILED DESCRIPTION:
Fresh tumor tissues and matched blood cells will be analyzed by large-panel (Berryoncology, lnc.) for multiple molecular biomarkers including mutations with sensitivity/resistance to targeted therapies, tumor mutational burden (TMB), microsatellite instability (MSI) status, etc., Therapeutic approach and outcome will be followed-up to inspect the clinical benefit by large-panel analysis. In addition, selected samples will be analyzed by WES to assess the correctness of TMB estimated by large-panel.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 or above, and gender unrestricted
* Individual with pathologically diagnosed lung cancer

Exclusion Criteria:

* Patients with concomitant other tumors
* Individual with severe cardiopulmonary insufficiency and hypoproteinemia
* Women who were pregnant and were during their lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in shanghai chest hospital
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through the whole study period, an average of 3 year
  PFS refers to the time from initial treatment to the time of disease progression or death
Tumor Mutational Burden (TMB) | halfway of the study, an average of 1.5 year
  TMB is defined as the total number of detected somatic mutation counts in coding regions per million bases

SECONDARY OUTCOMES:
Other biomarkers | halfway of the study, an average of 1.5 year
  The distribution and clinical application value of molecular biomarkers such as Neoantigen, MSI and LOH in Chinese lung cancer patients
Clonality | halfway of the study, an average of 1.5 year
  The tumor clonality in Chinese lung cancer patients
Overall survival (OS) | through the whole study period, an average of 3 year
  OS refers to the time from the patient entering into the group to the time of death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China